CLINICAL TRIAL: NCT04374799
Title: A Randomized Trial of Heparin vs Placebo in Patients Undergoing Cardiac Catheterization Via the Trans-radial Approach
Brief Title: Heparin vs Placebo for Cardiac Catheterization
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2102
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose heparin (Active Comparator): heparin (25 IU/Kg -maximal dose 3,000 IU)
  Interventions: Drug: Heparin
- High dose heparin (Active Comparator): heparin 50 IU/kg -maximal dose 5,000 IU
  Interventions: Drug: Heparin
- Placebo (Placebo Comparator): Normal saline 0.9%.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Heparin — two doses of heparin
  Arms: High dose heparin; Low dose heparin
Drug: Placebos — placebo
  Arms: Placebo

SUMMARY:
Patients undergoing cardiac catheterization will be randomized to 3 groups: no anticoagulant, low dose anticoagulant and high dose anticoagulant.

DETAILED DESCRIPTION:
Patients undergoing diagnostic cardiac catheterization via the trans-radial approach will be randomly allocated (1:1:1) to receive either low-dose UFH (25 IU/Kg -maximal dose 3,000 IU), high-dose UFH 50 IU/kg -maximal dose 5,000 IU) or N/S 0.9%. After 30 minutes, patients will undergo a gradual wrist band release. Hematoma and radial artery occlusion will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic cardiac catheterization; Small size sheath; patency of the ulno-palmar circulation

Exclusion Criteria:

abnormal ulno-palmar circulation; Prior radial artery thrombosis; Prior surgery close to the access site; Emergent cardiac catheterization; History of HIT or allergy to heparin; Patients requiring anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
hematoma | 1 hour
  >5 cm
radial artery occlusion | 1 hour
  by ultrasound

SECONDARY OUTCOMES:
access site bleeding | 1 hour
  any bleeding
non access site bleeding | 1 day
  bleeding not related to access site, such as gastrointestinal
access site complications | 1 day
  pseudoaneurysm, arteriovenous fistula
wrist band duration | 3 hours
  How long wrist band was on
time to discharge | 1 day
  when patient was able to leave the post procedure care area

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No